CLINICAL TRIAL: NCT06122545
Title: Chronic Migraine Prophylaxis: Comparative Study Between Ultrasound-Guided Greater Occipital Nerve Block and Medical Treatment
Brief Title: Chronic Migraine Prophylaxis: Ultrasound-Guided Greater Occipital Nerve Block Versus Medical Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sarah Zakaria Mohamed Elramady, Assistant Lecturer of Neurology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35459/4/22
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Greater Occipital Nerve Block; Medical Treatment; Chronic Migraine
MeSH Terms: interventions — Bupivacaine; onabotulinum toxin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greater Occipital Nerve Block (Experimental): Patients will receive greater occipital nerve block (GONB) either with local anesthetic (bupivacaine 0.5% 1.5 mL) or with onabotulinum toxin A injection.
  Ultrasound-guided Greater Occipital Nerve Block (GONB) will be performed to more accurately locate the nerve through searching for the occipital artery in the medial one-third of the superior nuchal line between the occipital tubercle and mastoid process and injection will be done medial to the artery
  Interventions: Procedure: Greater Occipital Nerve Block; Drug: bupivacaine or onabotulinum toxin A injection.
- Medical Treatment (Experimental): Patients who will receive medical treatment
  Interventions: Other: Medical Treatment

INTERVENTIONS:
Procedure: Greater Occipital Nerve Block — Patients will receive Greater Occipital Nerve Block (GONB) either with local anesthetic (bupivacaine 0.5% 1.5 mL) or with onabotulinum toxin A injection.
  Ultrasound-guided GONB will be performed to more accurately locate the nerve through searching for the occipital artery in the medial one-third of the superior nuchal line between the occipital tubercle and mastoid process and injection will be done medial to the artery
  Arms: Greater Occipital Nerve Block
Other: Medical Treatment — Patients who will receive medical treatment
  Arms: Medical Treatment
Drug: bupivacaine or onabotulinum toxin A injection. — bupivacaine 0.5% 1.5 mL) or with onabotulinum toxin A injection.
  Arms: Greater Occipital Nerve Block

SUMMARY:
The aim of this work is to assess the efficacy of ultrasound guided greater occipital nerve block either by local anesthetic or by botulinum toxin in comparison to medical treatment in prevention of chronic migraine.

DETAILED DESCRIPTION:
Primary headache disorders, particularly migraine and tension-type headache (TTH) are common worldwide and commonly result in widespread and substantial disability. Chronic migraine (CM) is defined as "headache occurring on 15 or more days per month for more than 3 months which has the features of migraine headache on at least 8 days per month".

The prevalence of CM in the general population is about 2%. It negatively affects emotional and family relationships, education, economic status, and general health. Migraine headaches might become quite severe and incapacitating for patients and management can be challenging even in experienced clinics.

Prophylactic interventions may include pharmacotherapy, behavioral therapy, physical therapy and other strategies. Management often requires the simultaneous use of these different therapeutic modalities. Once the headaches become refractory to conventional pharmacologic management minimally invasive techniques such as peripheral nerve blocks are feasible for pain relief and help to decrease the frequency of the attacks.

Preventive medications for chronic migraine treatment are less well studied than they are for episodic migraine. In addition, some trials evaluating treatment of chronic migraine are limited by one or more methodologic problems, such as small size, concomitant use of other prophylactic medications and/or lack of a specific headache diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old.
2. Both sexes.
3. Patients with chronic migraine.

Exclusion Criteria:

1. Age less than 18 years.
2. Patients with medication overuse headache.
3. Patients who had used acute pain medications within 24 hours prior to the study visit.
4. History of injury to the area of the GON.
5. Any prior adverse reactions to local anesthetics.
6. Patients with impaired sensation in the occipital area.
7. Any neurological or dermatological disease that may have affected skin sensation, bleeding tendency, any skull defect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
severity of headache | Follow up after 3 months
  severity of headache will be assessed by the total Migraine Disability Assessment (MIDAS) score used to define four grades of migraine-related disability with grade I for "little or no disability" (0-5); grade II for "mild disability" (6-10); grade III for "moderate disability" (11-20); and grade IV for "severe disability" (≥ 21).

SECONDARY OUTCOMES:
Reduction in headache days per month | Follow up after 3 months
  Reduction in headache days per month will be assessed by total Headache Impact Test 6 (HIT 6) score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent.
Migraine specific quality of life | Follow up after 3 months
  The total Migraine Disability Assessment (MIDAS) score range from 0 to 270 with the following disability classification criteria: (1) 0 to 5: slight or no disability, (2) 6 to 10: low levels of disability, (3) 11 to 20: moderate disability, and (4) 21 or above: severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.